CLINICAL TRIAL: NCT07240311
Title: Randomized Controlled Trial Evaluating AmblyoFix for the Treatment of Unilateral Amblyopia in Children, Teenagers and Young Adults Aged 8-35
Brief Title: Evaluation of AmblyoFix for the Treatment of Unilateral Amblyopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eyesight Electronics (Industry)
Collaborators: Nour Pajouhan Shargh Eye Specialist Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFX-RCT-IRN-2025
Record Dates: First submitted 2025-09-30; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- AmblyoFix (Experimental): Participants assigned to this arm will undergo binocular vision therapy using the AmblyoFix software on a laptop, in combination with red-blue anaglyph glasses. Prior to therapy initiation, a calibration process will be completed and validated by the study team to ensure device screen specifications meet protocol requirements. Treatment consists of interactive, gamified visual tasks designed to stimulate the amblyopic eye under binocular viewing conditions. Participants will complete 90 minutes of therapy per day, six days per week, for 24 weeks. The software includes adaptive difficulty adjustments, automated usage logging for compliance monitoring, and a daily lockout feature to prevent overuse. Parents/guardians will receive training materials to support session supervision and problem reporting.
  Interventions: Behavioral: AmblyoFix binocular digital therapy
- Patching (standard occlusion) (Active Comparator): Participants assigned to this arm will receive standard occlusion therapy consisting of patching the non-amblyopic eye for 2 hours per day, six days per week, over a 24-week period, while continuing to wear spectacles full time. Caregivers will be trained to correctly apply and monitor patching, maintain daily patching logs documenting hours patched and any issues, and identify signs of intolerance. Patching logs will be reviewed by investigators during scheduled follow-up visits.
  Interventions: Behavioral: Occlusion therapy (Patching)

INTERVENTIONS:
Behavioral: AmblyoFix binocular digital therapy — AmblyoFix is a binocular vision therapy delivered through specialized software on a laptop computer in combination with red-blue anaglyph glasses. The program uses interactive, gamified visual tasks designed to stimulate the amblyopic eye while maintaining binocular viewing conditions. Each participant undergoes a standardized calibration process to ensure screen specifications are validated before starting therapy. The prescribed regimen is 90 minutes per day, six days per week, for 24 weeks. The software incorporates adaptive difficulty adjustment, automated compliance logging with timestamped usage data, and a daily lockout feature to prevent overuse. Therapy adherence and performance are monitored remotely, and caregivers receive structured training materials to support session supervision and troubleshooting.
  Arms: AmblyoFix
Behavioral: Occlusion therapy (Patching) — Standard occlusion therapy involves patching of the non-amblyopic (fellow) eye to stimulate visual function in the amblyopic eye. Participants are prescribed patching for 2 hours per day, six days per week, over a 24-week treatment period, while continuing to wear their full-time spectacle correction. Caregivers are trained to correctly apply the patch, supervise adherence, and recognize signs of intolerance. Daily patching logs are maintained by caregivers to record hours patched and any issues encountered, and these logs are reviewed by investigators at scheduled follow-up visits.
  Arms: Patching (standard occlusion)

SUMMARY:
This is a prospective, randomized, parallel-group, assessor-masked, non-inferiority clinical trial designed to compare the efficacy, safety, and adherence of AmblyoFix binocular digital therapy with standard occlusion (patching) for the treatment of unilateral amblyopia in children and young adults aged 8 to 35 years. In the event that adequate recruitment within this age range is not feasible, the age range may be modified, subject to appropriate ethical approval and protocol amendment procedures.

A total of 86 participants will be enrolled (43 per arm). Eligible participants will be randomized in a 1:1 ratio to receive either AmblyoFix or patching, stratified by age group and amblyopia severity. Randomization will be implemented using the sealed opaque envelope method, with allocation concealment maintained through sequentially numbered, tamper-proof envelopes.

The primary outcome is the change in amblyopic-eye best-corrected visual acuity (BCVA, logMAR) from baseline to 24 weeks, assessed under standardized Snellen or ETDRS protocol. Secondary outcomes include adherence, safety, and patient-reported outcomes. An interim analysis will be performed at 12 weeks, with the option to stop the trial early if sufficient improvement in BCVA is demonstrated.

Participants and caregivers cannot be blinded due to the nature of the interventions; however, outcome assessors and statisticians will remain blinded to treatment allocation to minimize bias. Follow-up assessments will occur at baseline, 4, 8, 12, 16, 20 and 24 weeks, with no additional amblyopia treatment permitted during the study unless clinically required.

This trial aims to rigorously determine whether AmblyoFix is a safe, effective, and non-inferior alternative to standard patching, with the potential to improve adherence and acceptability in amblyopia therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-35 years.
* Unilateral amblyopia secondary to anisometropia, strabismus, or mixed.
* BCVA in amblyopic eye between 20/40-20/400 (0.3-1.3 logMAR); fellow eye ≥20/32 (≤0.2 logMAR).
* Interocular difference ≥2 lines (≥0.2 logMAR).
* Stable refractive correction for ≥16 weeks or <0.1 logMAR change across two visits ≥8 weeks apart.
* Cycloplegic refraction within 7 months meeting anisometropia criteria (e.g., hyperopia ≥+2.50 D).
* Access to a suitable home environment (laptop and internet) for AmblyoFix arm.
* Parent/guardian consent and child assent (8+ year olds).

Exclusion Criteria:

* Atropine use within 2 weeks before starting treatment
* Prior amblyopia treatment beyond refractive adaptation.
* Myopia >-6.00 D SE, previous ocular surgery, or other ocular pathology.
* Severe cognitive/developmental delay impeding compliance.
* History of light-induced seizures.
* Inability/unwillingness to comply with digital monitoring.
* Any condition compromising safety or trial integrity.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA in the amblyopic eye from baseline to Week 24 | From enrollment to the end of treatment at 24 Weeks
  The primary outcome of this trial is the change in best-corrected visual acuity (BCVA) in the amblyopic eye from baseline to week 24, measured in logMAR units using the Snellen or ETDRS protocol. This approach was selected for its clinical validity, reproducibility, and alignment with international standards in amblyopia trials, particularly for the study's target population of individuals aged 8-35 years. Visual acuity will be assessed monocularly under best optical correction, with the fellow eye occluded during testing. Certified, masked outcome assessors will conduct all measurements in standardized conditions to minimize bias, with testing procedures (including lighting, calibration, and display specifications) harmonized. Assessments will occur at baseline and at follow-up visits scheduled every 4 weeks during the 24-week intervention period, to monitor durability of treatment effects.

SECONDARY OUTCOMES:
Adherence to AmblyoFix | From enrollment to the end of treatment at 24 Weeks
  Adherence will be objectively measured through the AmblyoFix software's built-in time-tracking functions, which automatically record session frequency and duration. Adherence will be calculated as the total minutes of active use per week compared with the prescribed target duration. Mean weekly adherence will be derived over the 24-week treatment period.
  Unit of Measure:
  Total minutes of active use per week (minutes/week)
Adherence to occlusion therapy | From enrollment to Week 24
  Adherence will be monitored via parental reporting and a standardized compliance questionnaire administered at clinical visits. Parents will record the average number of hours per day that the prescribed occlusion therapy (eye patching) was completed. A mean reported adherence value will be calculated for each participant, expressed as the ratio of completed to prescribed hours per day.
  This questionnaire was developed for this study and has not been previously validated.
  Unit of Measure:
  Mean hours of occlusion per day (hours/day)
Safety of Amblyofix | From enrollment to the end of treatment at 24 Weeks
  Safety will be evaluated by recording all adverse events (AEs) and serious adverse events (SAEs) throughout the 24-week intervention period. Particular attention will be paid to ocular health, including reports of visual discomfort, diplopia, or any unexpected effects potentially related to digital therapy or occlusion. All safety data will be reviewed and summarized by the study investigators at each follow-up visit and at study completion.
  Unit of Measure:
  Number of participants with adverse events.
Patient Satisfaction | From enrollment to the end of treatment at 24 Weeks
  Patient satisfaction will be assessed using a custom 10-item questionnaire developed for this study. Each item is rated on a 5-point Likert scale (1 = very dissatisfied to 5 = very satisfied). The questionnaire evaluates four domains: acceptability, comfort, ease of use, and overall satisfaction. Scores will be averaged to produce a total satisfaction score, with higher values indicating greater satisfaction.
  This instrument was developed specifically for this trial and has not been previously validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nour Pajouhan Shargh Eye Specialist Clinic, Zahedan, Sistan & Balouchestan, Iran

IPD SHARING:
Plan to Share IPD: No